CLINICAL TRIAL: NCT05181930
Title: Nuclear Magnetic Resonance Spectroscopic Analysis of Urinary Metabolome in Sarcoidosis
Brief Title: Nuclear Magnetic Resonance Spectroscopic Analysis of Urinary Metabolome in Sarcoidosis (RMN-SARCURINES)
Acronym: RMN-SARCURINES
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01555-48
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2021-09

CONDITIONS: Sarcoidosis
Keywords: Sarcoidosis; Urinary; NMR spectroscopy; Metabolomic
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"Sarcoidosis is a systemic granulomatous disease of unknown cause(s).Determining disease activity is a major element in the treatment decision.

1H- Nuclear magnetic resonance (NMR) spectroscopy allows the identification of biomarkers in different pathologies and in particular in a pilot study of saliva of patients with sarcoidosis. Applications to sarcoidosis are still rare, having concerned only serum and saliva. In this context we hypothesize the existence of a difference in the metabolic products found in the urine of sarcoidosis patients with different degrees of activity and/or disease severity.

We designed an analysis of urinary metabolomics in sarcoidosis patient using NMR spectroscopy with multivariate statistical analysis, followed by metabolite identification and pathway analysis. "

DETAILED DESCRIPTION:
"Sarcoidosis is a systemic granulomatous disease of unknown cause(s) with an almost constant lung involvement. Clinical expression varies greatly in both evolution and severity. The activity of the disease is currently based on serum markers (elevation of angiotensin-converting enzyme) with poor sensitivity/specificity or on imaging techniques (18F-FDG PET-CT) which are more invasive and more expensive. Determining disease activity is a major element in the treatment decision.

The spectra of small molecules resulting from metabolism (metabolome/metabolomics) evaluated by spectrometry in different biological fluids (blood, saliva, urine) during different physiological or pathological conditions have been identified as promising biomarkers. 1H- Nuclear magnetic resonance (NMR) spectrometry allows the identification of biomarkers in different pathologies and in particular in a pilot study of saliva of patients with sarcoidosis. Applications to sarcoidosis are still rare having concerned only serum and saliva. The application of this method to the urinary metabolome has shown its effectiveness in other situations, for example in celiac disease.

In this context we hypothesize the existence of a difference in the metabolic products found in the urine of sarcoidosis patients with different degrees of activity and/or disease severity.

We designed an analysis of urinary metabolomics in sarcoidosis patient using NMR spectroscopy with multivariate statistical analysis, followed by metabolite identification and pathway analysis. "

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of sarcoidosis according to ATS / ERS / WASOG criteria.

Exclusion Criteria:

* Treatment (corticosteroids, plaquenil, immunosuppressants) within the last 6 months
* Patients with diabetes.
* Patient with long-term or recent drug treatment (e.g. antibiotics)
* Patients with a urinary tract infection or urinary lithiasis at the time of collection.
* Renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of sarcoidosis according to ATS / ERS / WASOG criteria consulting at the Pulmonary Department of the Avicenne University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Qualitative and quantitative analysis of NMR spectra of urine samples from a population of patients with sarcoidosis and comparison with an overall disease activity score | At inclusion
  NMR analysis on urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François BERNAUDIN, MD PhD, Principal Investigator — APHP
Locations (1):
- Hopital Avicenne,AP-HP, Bobigny, France

REFERENCES:
- [Background] Duchemann B, Triba MN, Guez D, Rzeznik M, Savarin P, Nunes H, Valeyre D, Bernaudin JF, Le Moyec L. Nuclear magnetic resonance spectroscopic analysis of salivary metabolome in sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 2016 Mar 29;33(1):10-6. PMID 27055831